CLINICAL TRIAL: NCT00924326
Title: An Assessment of the Safety and Feasibility of Administering T-Cells Expressing an Anti-CD19 Chimeric Antigen Receptor to Patients With B-Cell Lymphoma
Brief Title: CAR T Cell Receptor Immunotherapy for Patients With B-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 090082; 09-C-0082; NCT00862069 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Primary Mediastinal B-cell Lymphoma; Diffuse, Large B-cell Lymphoma; Diffuse Large B-Cell Lymphoma Transformed From Follicular Lymphoma; Mantle Cell
Keywords: B Cell Malignancies; T Cell Persistence; Immunotherapy; Cell Transfer; Leukemia; Chronic Lymphocytic Leukemia; CLL; Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- 1x10^9-1x10^10+ high dose Interleukin-2 (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + cryopreserved anti-CD19-CAR PBL
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Anti-cluster of differentiation 19 (CD19)-CAR PBL; Drug: Aldesleukin
- 1x10^9-1x10^10 + high dose Retreat (Experimental)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Anti-cluster of differentiation 19 (CD19)-CAR PBL; Drug: Aldesleukin
- 0.5x10^7 cells/kg (Experimental)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Anti-cluster of differentiation 19 (CD19)-CAR PBL
- 2.5x10^6 cells/kg (Experimental)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Anti-cluster of differentiation 19 (CD19)-CAR PBL
- 1.0x10^6 cells/kg (Experimental)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Anti-cluster of differentiation 19 (CD19)-CAR PBL
- 1.0x10^6 cells/kg (Reduced chemo) (Experimental)
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-CAR PBL; Drug: Fludarabine; Drug: Cyclophosphamide
- 2.0x10^6 cells/kg (Reduced chemo) (Experimental)
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-CAR PBL; Drug: Fludarabine; Drug: Cyclophosphamide
- 6.0x10^6 cells/kg (Reduced chemo) (Experimental)
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-CAR PBL; Drug: Fludarabine; Drug: Cyclophosphamide
- 2.0x10^6 cells/kg (Moderate chemo) (Experimental)
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-CAR PBL; Drug: Fludarabine; Drug: Cyclophosphamide
- 2.0x10^6 cells/kg (9-12 days culture) (Experimental)
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-CAR PBL; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Fludarabine — Days -5 to -1 (after administration of cyclophosphamide): 25 mg/m^2 intravenous (IV) over 30 minutes
  Other Names: Fludara
  Arms: 0.5x10^7 cells/kg; 1.0x10^6 cells/kg; 1x10^9-1x10^10 + high dose Retreat; 1x10^9-1x10^10+ high dose Interleukin-2; 2.5x10^6 cells/kg
Drug: Cyclophosphamide — Days -5 to -4: 60mg/kg intravenous (IV) over 60 minutes
  Other Names: Cytoxan
  Arms: 0.5x10^7 cells/kg; 1.0x10^6 cells/kg; 1x10^9-1x10^10 + high dose Retreat; 1x10^9-1x10^10+ high dose Interleukin-2; 2.5x10^6 cells/kg
Biological: Anti-cluster of differentiation 19 (CD19)-CAR PBL — Anti-cluster of differentiation 19 (CD19) chimeric antigen receptor (CAR) peripheral blood lymphocytes ( PBL).
  Day 0 (two to four days after the last dose of fludarabine); Cells will be infused via intravenous (IV) on the Patient Care Unit over 20-30 minutes.
Drug: Aldesleukin — Day 0: 720,000 IU/kg intravenously (IV) every 8 hours for a maximum of 15 doses.
  Other Names: Interleukin-2; IL-2
  Arms: 1x10^9-1x10^10 + high dose Retreat; 1x10^9-1x10^10+ high dose Interleukin-2
Drug: Fludarabine — Days -5 to -3 (after administration of cyclophosphamide): 30 mg/m^2 intravenous (IV) over 30 minutes
  Other Names: Fludara
  Arms: 1.0x10^6 cells/kg (Reduced chemo); 2.0x10^6 cells/kg (9-12 days culture); 2.0x10^6 cells/kg (Moderate chemo); 2.0x10^6 cells/kg (Reduced chemo); 6.0x10^6 cells/kg (Reduced chemo)
Drug: Cyclophosphamide — Days -5 to -3: 300mg/m^2 intravenous (IV) over 60 minutes
  Other Names: Cytoxan
  Arms: 1.0x10^6 cells/kg (Reduced chemo); 2.0x10^6 cells/kg (9-12 days culture); 2.0x10^6 cells/kg (Moderate chemo); 2.0x10^6 cells/kg (Reduced chemo); 6.0x10^6 cells/kg (Reduced chemo)

SUMMARY:
Background:

The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy for treating patients with B cell lymphomas or leukemias that involves taking white blood cells from the patient, growing them in the laboratory in large numbers, genetically modifying these specific cells with a type of virus (retrovirus) to attack only the tumor cells, and then giving the cells back to the patient. This type of therapy is called gene transfer. In this protocol, we are modifying the patient s white blood cells with a retrovirus that has the gene for anti-cluster of differentiation 19 (CD19) incorporated in the retrovirus.

Objective:

The purpose of this study is to determine a safe number of these cells to infuse and to see if these particular tumor-fighting cells (anti-CD19 cells) cause tumors to shrink.

Eligibility:

- Adults age 18-70 with B cell lymphomas or leukemias expressing the CD19 molecule.

Design:

Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed

Leukapheresis: If the patients meet all of the requirements for the study they will undergo leukapheresis to obtain white blood cells to make the anti-CD19 cells. Leukapheresis is a common procedure, which removes only the white blood cells from the patient.

Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy and the anti-CD19 cells. They will stay in the hospital for about 4 weeks for the treatment.

Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits will take up to 2 days.

DETAILED DESCRIPTION:
BACKGROUND:

* We have constructed a retroviral vector that encodes an anti-cluster of differentiation 19 (CD19) chimeric antigen receptor (CAR) that recognizes the CD19 antigen. This chimeric receptor also contains the signaling domains of cluster of differentiation 28 (CD28) and cluster of differentiation 3 (CD3)-zeta. The retroviral vector can be used to mediate genetic transfer of this CAR to T cells with high efficiency (> 50%) without the need to perform any selection.
* In co-cultures with CD19-expressing target cells, anti-CD19-CAR-transduced T-cells secreted significant amounts of interferon gamma (IFN-y) and interleukin 2 (IL-2).
* We have developed a process for cryopreserving the cell product which may lead to the ability for this product to be manufactured at a central location and shipped to other institutions for treatment of a broader patient population

OBJECTIVE:

- Primary objective:

--With the approval of amendment S, to determine the safety and feasibility of the administration of cryopreserved anti-CD19-CAR engineered peripheral blood lymphocytes with a non-myeloablative conditioning regimen in patients with Bcell lymphomas.

ELIGIBILITY:

Patients of 18 years of age or older must:

* Have a CD19-expressing B-cell lymphoma
* Be a non-responder to, or recurred after one or more standard chemotherapy-containing regimens for their malignancy
* Currently require treatment due to progressive malignancy
* Be deemed to be incurable by standard therapy

Patients may not have:

* A history of allogeneic stem cell transplantation
* Central nervous system (CNS) disease

DESIGN:

* Peripheral blood mononuclear cells (PBMC) obtained by leukapheresis (approximately 5.0x 10^9 cells) will be cultured in the presence of anti-CD3 (muromonab-CD3 (OKT3)) and aldesleukin in order to stimulate T-cell proliferation.
* Transduction is initiated by exposure of approximately 1.0x 10^8 to 5.0x 10^8 cells to retroviral vector supernatant containing the anti-CD19 CAR.
* With the approval of Amendment S, patients will receive fludarabine and cyclophosphamide chemotherapy (NMA) for lymphodepletion, followed by cryopreserved anti-CD19-CAR-transduced T-cells.
* Patients will be followed until disease progression.
* Patients who have responded to treatment and then progress may receive one retreatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patient must have a cluster of differentiation 19 (CD19)-expressing B-cell lymphoma. Patients with diffuse large B-cell lymphoma, primary mediastinal B-cell lymphoma, and diffuse large B-cell lymphoma transformed from follicular lymphoma must have measurable disease after at least two prior chemotherapy regimens one of which must have contained doxorubicin and rituximab.
  2. Confirmation of diagnosis of B-cell malignancy and positivity for CD19 confirmed by the Laboratory of Pathology of the National Cancer Institute (NCI). The choice of whether to use flow cytometry or immunohistochemistry will be determined by what is the most easily available tissue sample in each patient. Immunohistochemistry will be used for lymph node biopsies, flow cytometry will be used for peripheral blood, fine needle aspirates and bone marrow samples.
  3. Patients must have indications for treatment for their B-cell malignancy at the time of enrollment on this trial.
  4. Greater than or equal to 18 years of age and less than or equal to age 70.
  5. Willing to sign a durable power of attorney.
  6. Able to understand and sign the Informed Consent Document.
  7. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  8. Life expectancy of greater than three months.
  9. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for four months after treatment.
  10. Women of child bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
  11. Serology:

      * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.).
      * Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative. If hepatitis C antibody test is positive. Then patients must be tested for the presence of antigen by reverse transcription-polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
  12. Hematology:

      * Absolute neutrophil count greater than or equal to 1000/mm^3 without the support of filgrastim.
      * Platelet count greater than or equal to 50,000/mm^3.
      * Hemoglobin greater than 8.0 g/dl.
      * Lymphocyte count less than or equal to 4,000/ mm^3
  13. Chemistry:

      * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 5 times the upper limit of normal.
      * Serum creatinine less than or equal to 1.6 mg/dl
      * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl
  14. More than three weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patient toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
  15. Normal cardiac ejection fraction and no evidence of pericardial effusion as determined by an echocardiogram.

EXCLUSION CRITERIA:

1. Patients that require urgent therapy due to tumor mass effects such as bowel obstruction or blood vessel compression.
2. Patients that have active hemolytic anemia.
3. Patients with active brain metastases, or with a history of any central nervous system (CNS) metastases or cerebrospinal fluid malignant cells.

   Note: patients who are asymptomatic but are found to have malignant cells in the cerebrospinal fluid (CSF) on lumbar puncture prior to treatment will be considered eligible.
4. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
5. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
6. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
7. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
8. Concurrent systemic steroid therapy.
9. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
10. History of allogeneic stem cell transplantation
11. Patients with cardiac atrial or cardiac ventricular lymphoma involvement.

Screening Evaluation:

Within 4 weeks prior to starting the chemotherapy regimen:

1. Complete history and physical examination, including, weight and vital signs, noting in detail the exact size and location of any lesions that exist. (Note: patient history may be obtained within 8 weeks.)
2. Chest x-ray
3. Electrocardiography (EKG)
4. Baseline computed tomography (CT) of the chest, abdomen and pelvis, positron emission tomography (PET) scan, and brain magnetic resonance imaging (MRI) to evaluate the status of disease. Additional scans and x-rays may be performed if clinically indicated based on patient signs and symptoms.
5. HIV antibody titer and Hepatitis B surface antigen (HbsAG) determination, and anti HCV, (Note: May be performed within 3 months of the chemotherapy start date).
6. Anti cytomegalovirus (CMV) antibody titer, herpes simplex virus (HSV) serology, and Epstein-Barr virus (EBV) panel (Note: patients who are known to be positive for any of the above do not need to be retested; may be performed within 3 months of chemotherapy start date)
7. Patients with a left ventricular ejection fraction (LVEF) of less than or equal to 55% will not proceed to treatment (Note: may be performed within 8 weeks of treatment).
8. Cluster of differentiation 19 (CD19) staining of malignant cells by immunohistochemistry or flow cytometry (testing is permitted to be conducted at any time prior to this point).
9. All patients must have a T cells, B cells, and natural killer cells (TBNK) for Peripheral blood cluster of differentiation 3 (CD3) count and CD19#.
10. Patients with a history of leptomeningeal disease, or signs/symptoms suggestive of leptomeningeal involvement, or with symptoms of central nervous system malignancy such as new onset severe headaches, neck stiffness, or any focal neurologic findings on physical exam will have lumbar puncture for examination of cerebral spinal fluid.
11. Patients may undergo lumbar puncture (LP) for flow cytometry of the CSF in order to assess the presence of CD19 positive lymphocytes for potential correlation with neurologic toxicity. Patients who have no neurologic symptoms at the time of LP will be eligible for enrollment regardless of the results of the flow cytometry.

    Within 14 days prior to starting the chemotherapy regimen:
12. Chem 20: (Sodium (Na), Potassium (K), Chloride (Cl), Total carbon dioxide (CO2) (bicarbonate), Creatinine, Glucose, Urea nitrogen (BUN), Albumin, Calcium total, Magnesium total (Mg), Inorganic Phosphorus, Alkaline Phosphatase, ALT/glutamic pyruvic transaminase (GPT), AST/glutamic oxaloacetic (GOT), Total Bilirubin, Direct Bilirubin, lactate hydrogenase (LD), Total Protein, Total creatine kinase (CK), Uric Acid)
13. Thyroid panel
14. Complete blood count (CBC) with differential and platelet count
15. Prothrombin time (PT)/partial thromboplastin time (PTT)
16. Urinalysis and culture, if indicated

    Within 7 days prior to starting the chemotherapy regimen:
17. Beta-human chorionic gonadotropin (βHCG) pregnancy test (serum or urine) on all women of child-bearing potential
18. ECOG performance status of 0 or 1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-02-17 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2021-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kochenderfer JN, Rosenberg SA. Treating B-cell cancer with T cells expressing anti-CD19 chimeric antigen receptors. Nat Rev Clin Oncol. 2013 May;10(5):267-76. doi: 10.1038/nrclinonc.2013.46. Epub 2013 Apr 2. PMID 23546520
- [Result] Kochenderfer JN, Dudley ME, Carpenter RO, Kassim SH, Rose JJ, Telford WG, Hakim FT, Halverson DC, Fowler DH, Hardy NM, Mato AR, Hickstein DD, Gea-Banacloche JC, Pavletic SZ, Sportes C, Maric I, Feldman SA, Hansen BG, Wilder JS, Blacklock-Schuver B, Jena B, Bishop MR, Gress RE, Rosenberg SA. Donor-derived CD19-targeted T cells cause regression of malignancy persisting after allogeneic hematopoietic stem cell transplantation. Blood. 2013 Dec 12;122(25):4129-39. doi: 10.1182/blood-2013-08-519413. Epub 2013 Sep 20. PMID 24055823
- [Result] James N. Kochenderfer, M.D., Mark E. Dudley, Ph.D., Sadik H. Kassim, Ph.D., Robert O. Carpenter, James C. Yang, MD, Giao Q. Phan, MD, Marybeth S. Hughes, MD, Richard M. Sherry, MD, Steven Feldman, Ph.D., David Spaner, MD, PhD, Debbie-Ann N. Nathan, RN, Kathleen E. Morton, RN, Mary Ann Toomey, RN, and Steven A. Rosenberg, M.D., Ph.D. Effective Treatment of Chemotherapy-Refractory Diffuse Large B-Cell Lymphoma with Autologous T Cells Genetically-Engineered to Express an Anti-CD19 Chimeric Antigen Receptor. Oral Abstract Presentation 12-8-13 in New Orleans, LA at the American Society of Hematology annual meeting. Blood Annual Meeting abstract 2013. 122:168.
- [Result] Kochenderfer JN, Dudley ME, Kassim SH, Somerville RP, Carpenter RO, Stetler-Stevenson M, Yang JC, Phan GQ, Hughes MS, Sherry RM, Raffeld M, Feldman S, Lu L, Li YF, Ngo LT, Goy A, Feldman T, Spaner DE, Wang ML, Chen CC, Kranick SM, Nath A, Nathan DA, Morton KE, Toomey MA, Rosenberg SA. Chemotherapy-refractory diffuse large B-cell lymphoma and indolent B-cell malignancies can be effectively treated with autologous T cells expressing an anti-CD19 chimeric antigen receptor. J Clin Oncol. 2015 Feb 20;33(6):540-9. doi: 10.1200/JCO.2014.56.2025. Epub 2014 Aug 25. PMID 25154820
- [Result] Kochenderfer JN, Somerville RPT, Lu T, Shi V, Bot A, Rossi J, Xue A, Goff SL, Yang JC, Sherry RM, Klebanoff CA, Kammula US, Sherman M, Perez A, Yuan CM, Feldman T, Friedberg JW, Roschewski MJ, Feldman SA, McIntyre L, Toomey MA, Rosenberg SA. Lymphoma Remissions Caused by Anti-CD19 Chimeric Antigen Receptor T Cells Are Associated With High Serum Interleukin-15 Levels. J Clin Oncol. 2017 Jun 1;35(16):1803-1813. doi: 10.1200/JCO.2016.71.3024. Epub 2017 Mar 14. PMID 28291388
- [Result] James N. Kochenderfer, Mark E. Dudley, Robert O. Carpenter, Sadik H. Kassim, Jeremy J. Rose, William G. Telford, Frances T. Hakim, David C. Halverson, Daniel H. Fowler, Nancy M. Hardy, Anthony R. Mato, Dennis D. Hickstein, Juan C. Gea-Banacloche, Steven Z. Pavletic, Claude Sportes, Irina Maric, Steven A. Feldman, Brenna G. Hansen, Jennifer S. Wilder, Bazetta Blacklock-Schuver, Bipulendu Jena, Michael R. Bishop, Steven A. Rosenberg*, Ronald E. Gress* (co-senior authors). Donor-derived anti-CD19 chimeric-antigen-receptor-expressing T cells cause regression of malignancy persisting after allogeneic hematopoietic stem cell transplantation. Oral Abstract Presentation 12-8-13 in New Orleans, LA at the American Society of Hematology annual meeting. Blood Annual Meeting abstracts 2013. 122:151.
- [Result] Kochenderfer, J.N., Somerville, R., Lu, T., Shi, V., Yang, J.C., Sherry, R., Klebanoff, C., Kammula, U.S., Goff, S.L., Bot, A., Rossi, J., Sherman, M., Perez, A., Xue, A., Feldman, T.A., Friedberg, J.W., Roschewski, M.J., Feldman, S., McIntyre, L., Rosenberg, S.A. Anti-CD19 Chimeric Antigen Receptor T cells Preceded by Low-Dose Chemotherapy to Induce Remissions of Advanced Lymphoma. 2016 ASCO Annual Meeting. J Clin Oncol 34, 2016 (suppl; abstr LBA3010).
- [Result] Kochenderfer JN, Somerville RPT, Lu T, Yang JC, Sherry RM, Feldman SA, McIntyre L, Bot A, Rossi J, Lam N, Rosenberg SA. Long-Duration Complete Remissions of Diffuse Large B Cell Lymphoma after Anti-CD19 Chimeric Antigen Receptor T Cell Therapy. Mol Ther. 2017 Oct 4;25(10):2245-2253. doi: 10.1016/j.ymthe.2017.07.004. Epub 2017 Jul 13. PMID 28803861
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Cappell KM, Sherry RM, Yang JC, Goff SL, Vanasse DA, McIntyre L, Rosenberg SA, Kochenderfer JN. Long-Term Follow-Up of Anti-CD19 Chimeric Antigen Receptor T-Cell Therapy. J Clin Oncol. 2020 Nov 10;38(32):3805-3815. doi: 10.1200/JCO.20.01467. Epub 2020 Oct 6. PMID 33021872
- [Derived] Rossi J, Paczkowski P, Shen YW, Morse K, Flynn B, Kaiser A, Ng C, Gallatin K, Cain T, Fan R, Mackay S, Heath JR, Rosenberg SA, Kochenderfer JN, Zhou J, Bot A. Preinfusion polyfunctional anti-CD19 chimeric antigen receptor T cells are associated with clinical outcomes in NHL. Blood. 2018 Aug 23;132(8):804-814. doi: 10.1182/blood-2018-01-828343. Epub 2018 Jun 12. PMID 29895668
- [Derived] Kochenderfer JN, Dudley ME, Feldman SA, Wilson WH, Spaner DE, Maric I, Stetler-Stevenson M, Phan GQ, Hughes MS, Sherry RM, Yang JC, Kammula US, Devillier L, Carpenter R, Nathan DA, Morgan RA, Laurencot C, Rosenberg SA. B-cell depletion and remissions of malignancy along with cytokine-associated toxicity in a clinical trial of anti-CD19 chimeric-antigen-receptor-transduced T cells. Blood. 2012 Mar 22;119(12):2709-20. doi: 10.1182/blood-2011-10-384388. Epub 2011 Dec 8. PMID 22160384
- [Derived] Kochenderfer JN, Wilson WH, Janik JE, Dudley ME, Stetler-Stevenson M, Feldman SA, Maric I, Raffeld M, Nathan DA, Lanier BJ, Morgan RA, Rosenberg SA. Eradication of B-lineage cells and regression of lymphoma in a patient treated with autologous T cells genetically engineered to recognize CD19. Blood. 2010 Nov 18;116(20):4099-102. doi: 10.1182/blood-2010-04-281931. Epub 2010 Jul 28. PMID 20668228
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0082.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients treated in arm 1 (1x10e9-1x10e10 cells/kg + high dose IL2) had disease progression and were then retreated in Period 2 (1x10e9-1x10e10 cells/kg + high dose IL2).
Groups:
- 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2: Cyclophosphamide (Days -5 to -4): 60mg/kg intravenous (IV) over 60 minutes
  Fludarabine (Days -5 to -1 after administration of cyclophosphamide): 25 mg/m^2 intravenous (IV) over 30 minutes
  Anti-CD19 CAR PBL (Day 0 two to four days after the last dose of fludarabine); Cells will be infused via intravenous (IV) on the Patient Care Unit over 20-30 minutes.
  Aldesleukin (Day 0): 720,000 IU/kg intravenously (IV) every 8 hours for a maximum of 15 doses.
- 0.5x10^7 Cells/kg; 2.5x10^6 Cells/kg; 1.0x10^6 Cells/kg: Cyclophosphamide (Days -5 to -4): 60mg/kg intravenous (IV) over 60 minutes
  Fludarabine (Days -5 to -1 after administration of cyclophosphamide): 25 mg/m^2 intravenous (IV) over 30 minutes
  Anti-CD19 CAR PBL (Day 0 two to four days after the last dose of fludarabine); Cells will be infused via intravenous (IV) on the Patient Care Unit over 20-30 minutes.
- 1.0x10^6 Cells/kg (Reduced Chemo); 2.0x10^6 Cells/kg (Reduced Chemo); 6.0x10^6 Cells/kg (Reduced Chemo); 2.0x10^6 Cells/kg (Moderate Chemo); 2.0x10^6 Cells/kg (9-12 Days Culture): Cyclophosphamide (Days -5 to -3): 300mg/m^2 intravenous (IV) over 60 minutes
  Fludarabine (Days -5 to -3: after administration of cyclophosphamide): 30 mg/m^2 intravenous (IV) over 30 minutes
  Anti-CD19 CAR PBL (Day 0, two to four days after the last dose of fludarabine): Cells will be infused via intravenous (IV) on the Patient Care Unit over 20-30 minutes.
Period: Dose Administration
Arm/Group | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 | 0.5x10^7 Cells/kg | 2.5x10^6 Cells/kg | 1.0x10^6 Cells/kg | 1.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Reduced Chemo) | 6.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Moderate Chemo) | 2.0x10^6 Cells/kg (9-12 Days Culture)
Started | 8 | 2 | 5 | 6 | 7 | 10 | 1 | 2 | 2
Completed | 8 | 2 | 5 | 6 | 7 | 10 | 1 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 1x10^9-1x10^10 + High Dose Retreat
Arm/Group | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 | 0.5x10^7 Cells/kg | 2.5x10^6 Cells/kg | 1.0x10^6 Cells/kg | 1.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Reduced Chemo) | 6.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Moderate Chemo) | 2.0x10^6 Cells/kg (9-12 Days Culture)
Started | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 0.5x10^7 Cells/kg: Cyclophosphamide (Days -5 to -4): 60mg/kg intravenous (IV) over 60 minutes
  Fludarabine (Days -5 to -1 after administration of cyclophosphamide): 25 mg/m^2 intravenous (IV) over 30 minutes
  Anti-CD19 CAR PBL (Day 0 two to four days after the last dose of fludarabine); Cells will be infused via intravenous (IV) on the Patient Care Unit over 20-30 minutes.
  Aldesleukin (Day 0): 720,000 IU/kg intravenously (IV) every 8 hours for a maximum of 15 doses.
- Total: Total of all reporting groups
Arm/Group | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 | 0.5x10^7 Cells/kg | 2.5x10^6 Cells/kg | 1.0x10^6 Cells/kg | 1.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Reduced Chemo) | 6.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Moderate Chemo) | 2.0x10^6 Cells/kg (9-12 Days Culture) | Total
Number analyzed (Participants) | 8 | 2 | 5 | 6 | 7 | 10 | 1 | 2 | 2 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 2 | 5 | 5 | 5 | 8 | 1 | 2 | 1 | 37
  >=65 years | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (5.7) | 52.0 (12.7) | 40.4 (6.8) | 58.0 (8.6) | 55.0 (13.7) | 52.1 (15.2) | 40.0 | 51.5 (2.1) | 58.5 (10.6) | 52.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 4 | 0 | 2 | 0 | 0 | 1 | 10
  Male | 8 | 1 | 3 | 2 | 7 | 8 | 1 | 2 | 1 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 8 | 2 | 4 | 6 | 7 | 9 | 1 | 2 | 2 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 8 | 2 | 4 | 5 | 6 | 10 | 1 | 2 | 2 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 2 | 5 | 6 | 7 | 10 | 1 | 2 | 2 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response Assessed by the Response Criteria for Malignant Lymphoma
Description: Participants were assessed by the Response Criteria for Malignant Lymphoma. Complete Remission (CR) is complete disappearance of all detectable evidence of disease and disease-related symptoms if present before therapy. Partial Remission (PR) requires ≥50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses; no increase in size of nodes, liver or spleen and no new sites of disease. Progressive disease (PD) is defined by ≥50% increase from nadir in the sum of the products of at least two lymph nodes, or if a single node is involved at least a 50% increase in the product of the diameters of this one node; and appearance of a new lesion greater than 1.5 cm in any axis even if other lesions are decreasing in size. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Scans performed at 6 weeks, 12 weeks and every 3-6 months for approximately 2 years
Population: 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 Retreat Arm/Group: "3 participants in group 1 (1x10e9-1x10e10 cells/kg + high-dose IL2)) initially responded but were then retreated in group 2 after progression."
Measure: Count of Participants; unit: Participants
Groups:
- 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 Retreat: Cyclophosphamide (Days -5 to -4): 60mg/kg intravenous (IV) over 60 minutes
  Fludarabine (Days -5 to -1 after administration of cyclophosphamide): 25 mg/m^2 intravenous (IV) over 30 minutes
  Anti-CD19 CAR PBL (Day 0 two to four days after the last dose of fludarabine); Cells will be infused via intravenous (IV) on the Patient Care Unit over 20-30 minutes.
  Aldesleukin (Day 0): 720,000 IU/kg intravenously (IV) every 8 hours for a maximum of 15 doses.
Arm/Group | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 Retreat | 0.5x10^7 Cells/kg | 2.5x10^6 Cells/kg | 1.0x10^6 Cells/kg | 1.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Reduced Chemo) | 6.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Moderate Chemo) | 2.0x10^6 Cells/kg (9-12 Days Culture)
Number analyzed (Participants) | 8 | 3 | 2 | 5 | 6 | 7 | 10 | 1 | 2 | 2
Participants
  Complete Remission | 2 | 3 | 2 | 3 | 3 | 2 | 6 | 0 | 2 | 2
  Partial Remission | 4 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0
  Stable Disease | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Progressive Disease | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 0
  Not Evaluable | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0).
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 101 months and 17 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 Retreat | 0.5x10^7 Cells/kg | 2.5x10^6 Cells/kg | 1.0x10^6 Cells/kg | 1.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Reduced Chemo) | 6.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Moderate Chemo) | 2.0x10^6 Cells/kg (9-12 Days Culture)
Number analyzed (Participants) | 8 | 3 | 2 | 5 | 6 | 7 | 10 | 1 | 2 | 2
Participants | 8 | 1 | 2 | 5 | 6 | 7 | 10 | 1 | 2 | 2

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 101 months and 17 days.
Arm/Group | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 Retreat | 0.5x10^7 Cells/kg | 2.5x10^6 Cells/kg | 1.0x10^6 Cells/kg | 1.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Reduced Chemo) | 6.0x10^6 Cells/kg (Reduced Chemo) | 2.0x10^6 Cells/kg (Moderate Chemo) | 2.0x10^6 Cells/kg (9-12 Days Culture)
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/3 | 0/2 | 1/5 | 0/6 | 0/7 | 0/10 | 0/1 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 7/8 | 1/3 | 2/2 | 3/5 | 2/6 | 2/7 | 7/10 | 1/1 | 2/2 | 2/2
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3 | 2/2 | 5/5 | 6/6 | 7/7 | 10/10 | 1/1 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 (N=8) | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 Retreat (N=3) | 0.5x10^7 Cells/kg (N=2) | 2.5x10^6 Cells/kg (N=5) | 1.0x10^6 Cells/kg (N=6) | 1.0x10^6 Cells/kg (Reduced Chemo) (N=7) | 2.0x10^6 Cells/kg (Reduced Chemo) (N=10) | 6.0x10^6 Cells/kg (Reduced Chemo) (N=1) | 2.0x10^6 Cells/kg (Moderate Chemo) (N=2) | 2.0x10^6 Cells/kg (9-12 Days Culture) (N=2)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Abdomen NOS
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Valvular heart disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Neuropathy: cranial::CN VII Motor-face; Sensory-taste (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death not associated with CTCAE term (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyramidal tract dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — (e.g., increased tone, hyperreflexia, positive Babinski, decreased fine motor coordination)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 2 (3) | 2 (2)
Syndromes - Other (Myelodysplastic syndrome) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (incoordination) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Incontinence, urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Mood alteration::Agitation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 (N=8) | 1x10^9-1x10^10 Cells/kg + High-dose Interleukin-2 Retreat (N=3) | 0.5x10^7 Cells/kg (N=2) | 2.5x10^6 Cells/kg (N=5) | 1.0x10^6 Cells/kg (N=6) | 1.0x10^6 Cells/kg (Reduced Chemo) (N=7) | 2.0x10^6 Cells/kg (Reduced Chemo) (N=10) | 6.0x10^6 Cells/kg (Reduced Chemo) (N=1) | 2.0x10^6 Cells/kg (Moderate Chemo) (N=2) | 2.0x10^6 Cells/kg (9-12 Days Culture) (N=2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute vascular leak syndrome (Vascular disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood/Bone Marrow - Other (Hypogammaglobulinemia (IG A)) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood/Bone Marrow - Other (Hypogammaglobulinemia (IGG)) (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood/Bone Marrow - Other (Hypogammaglobulinemia (IG M)) (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (4) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 5 (5) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 8 (8) | 1 (1) | 1 (1) | 2 (2)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/Bleeding - Other (Subconjunctival hemorrhages) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Congenital, familial and genetic disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Colon
Infection with normal ANC or Grade 1 or 2 neutrophils::External ear (otitis externa) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Middle ear (otitis media) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Nerve-peripheral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Paranasal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 3 or 4 neutrophils::Blood (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Wound
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal nerve dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 8 (9) | 3 (3) | 2 (3) | 5 (5) | 6 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 8 (8) | 3 (5) | 2 (2) | 5 (5) | 6 (6) | 7 (7) | 10 (10) | 1 (1) | 1 (1) | 2 (2)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood alteration::Agitation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood alteration::Anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood alteration::Depression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: cranial: CN III Pupil, upper eyelid, extra ocular movements (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 8 (9) | 3 (3) | 2 (3) | 5 (5) | 5 (5) | 7 (7) | 9 (9) | 0 (0) | 1 (1) | 2 (2)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (3) | 1 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 8 (8) | 3 (3) | 2 (2) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (low urine output) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (Oliguria) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT00924326/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT00924326/ICF_002.pdf